CLINICAL TRIAL: NCT02539992
Title: A Prospective, Randomized, Multi-centre Study of the Triathlon Cruciate Retaining Total Knee System Using ShapeMatch Cutting Guides
Brief Title: ShapeMatch Cutting Guide Functional Outcomes Study
Acronym: ShapeMatch
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Product discontinued in November 2014
Sponsor: Stryker Orthopaedics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: K-S-045
Record Dates: First submitted 2015-09-01; First posted 2015-09-03 (Estimated); Results first posted 2016-05-16 (Estimated); Last update posted 2024-02-22 (Actual); Status verified 2024-02

CONDITIONS: Arthroplasty, Replacement, Knee

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Triathlon® CR/Kinematic Alignment (Active Comparator): Receive the Triathlon® Cruciate Retaining Total Knee System (Triathlon® CR) in a procedure using patient-specific cutting guides to reproduce the natural kinematic alignment of the knee.
  Interventions: Device: Triathlon® CR/Kinematic Alignment
- Triathlon® CR/Neutral Overall Limb Alignment (Active Comparator): Receive the Triathlon® CR device in a procedure using patient-specific cutting guides modified to provide neutral overall limb alignment of the knee.
  Interventions: Device: Triathlon® CR/Neutral Overall Limb Alignment
- Triathlon® CR/Conventional Limb Alignment (Active Comparator): Receive the Triathlon® CR device in a procedure using traditional instrumentation intended to achieve a neutral overall limb alignment of the knee.
  Interventions: Device: Triathlon® CR/Conventional Limb Alignment

INTERVENTIONS:
Device: Triathlon® CR/Kinematic Alignment — Total knee replacement using patient-specific cutting guides
  Arms: Triathlon® CR/Kinematic Alignment
Device: Triathlon® CR/Neutral Overall Limb Alignment — Total knee replacement using patient-specific cutting guides
  Arms: Triathlon® CR/Neutral Overall Limb Alignment
Device: Triathlon® CR/Conventional Limb Alignment — Total knee replacement using traditional instrumentation
  Arms: Triathlon® CR/Conventional Limb Alignment

SUMMARY:
Randomized evaluation of the ShapeMatch Cutting Guide for primary total knee replacement (TKR) in a consecutive series of patients who meet the eligibility criteria.

DETAILED DESCRIPTION:
This study will be a prospective, randomized evaluation of the ShapeMatch Cutting Guide for primary total knee replacement (TKR) in a consecutive series of patients who meet the eligibility criteria. Forty-eight cases enrolled will receive the Triathlon® Cruciate Retaining Total Knee System (Triathlon® CR) in a procedure using patient-specific cutting guides to reproduce the natural kinematic alignment of the knee. Another forty-eight cases enrolled will receive the Triathlon® CR device in a procedure using patient-specific cutting guides modified to provide neutral overall limb alignment of the knee. And the last forty-eight cases will receive the Triathlon® CR device in a procedure using traditional instrumentation intended to achieve a neutral overall limb alignment.

ELIGIBILITY:
Inclusion Criteria:

1. Patient has signed an ethic commission approved study specific Informed Patient Consent Form.
2. Patient is a male or non-pregnant female age 18 years or older at time of study device implantation.
3. Patient has primary diagnosis of Non-Inflammatory Degenerative Joint Disease (NIDJD).
4. Patient is a candidate for a primary total knee replacement.
5. Patient is willing and able to comply with postoperative scheduled clinical and radiographic evaluations and rehabilitation.

Exclusion Criteria:

1. Patient has a Body Mass Index (BMI) ≥ 40.
2. Patient age ≥ 80.
3. Patient has a varus or valgus deformity greater than 10 degree or flexion contracture greater than 20 degree.
4. Patient has an active or suspected latent infection in or about the affected knee joint at time of study device implantation.
5. Patient has received any orthopaedic surgical intervention to the lower extremities within the past year or is expected to require any orthopaedic surgical intervention to the lower extremities, other than the TKR to be enrolled in this study, within the next year.
6. Patient requires bilateral total knee replacements, or has a history of contralateral partial or total knee replacement.
7. Patient has any implanted device that would be incompatible with MRI procedures.
8. Patient has chronic heart failure (NYHA Stage ≥ 2)
9. Patient has a neuromuscular or neurosensory deficiency, which limits the ability to evaluate the safety and efficacy of the device.
10. Patient is diagnosed with a systemic disease (e.g. Lupus Erythematosus) or a metabolic disorder (e.g. Paget"s Disease) leading to progressive bone deterioration.
11. Patient is immunologically suppressed or receiving steroids in excess of normal physiological requirements (e.g. > 30 days).
12. Patient requires revision surgery of a previously implanted total knee replacement or knee fusion to the affected joint.
13. Patient has a known sensitivity to device materials.
14. Patient is a prisoner.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2012-05; Primary Completion 2015-05 (Actual); Study Completion 2015-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Fabio Catani, Prof., Principal Investigator — Azienada Ospedaliero-Universitaria di Modena
Locations (4):
- Medizinische Hochschule Hannover, Hanover, Lower Saxony, Germany
- Italy (2):
  - Istituto Ortopedico Rizzoli, Bologna, Emilia-Romagna
  - Azienada Ospedaliero-Universitaria di Modena, Modena
- Royal Devon and Exeter NHS Foundation Trust, Exeter, Devon, United Kingdom

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 56 patients have been screened for study participation. No patient withdrew his/her informed consent.
Pre-assignment Details: 12/56 patients received another procedure. Therefore 44 patients were enrolled in 4 centers.
Period: Overall Study
Arm/Group | Triathlon® CR/Kinematic Alignment | Triathlon® CR/Neutral Overall Limb Alignment | Triathlon® CR/Conventional Limb Alignment
Started | 15 | 11 | 18
Completed | 15 | 7 | 14
Not Completed | 0 | 4 | 4

BASELINE CHARACTERISTICS:
Population: Forty-four (44) patients were enrolled over an 11 month period in a randomized manner in 4 centers.
Groups:
- Total: Total of all reporting groups
Arm/Group | Triathlon® CR/Kinematic Alignment | Triathlon® CR/Neutral Overall Limb Alignment | Triathlon® CR/Conventional Limb Alignment | Total
Number analyzed (Participants) | 15 | 11 | 18 | 44
Age, Continuous [Mean (Standard Deviation); unit: years] | 69 (5.8) | 67 (9.3) | 70 (4.8) | 69 (6.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 7 | 10 | 26
  Male | 6 | 4 | 8 | 18
Region of Enrollment [Number; unit: participants]
  Italy | 11 | 7 | 12 | 30
  United Kingdom | 1 | 1 | 4 | 6
  Germany | 3 | 3 | 2 | 8

OUTCOME MEASURES:

1. Primary Outcome: Assessment of Better Functional Performance of Total Knee Replacement (TKR) Using a Kinematic Aligned ShapeMatch Cutting Guide by Means of Fluoroscopy.
Description: To demonstrate by means of fluoroscopy that TKR's performed using a kinematic aligned ShapeMatch Cutting Guide provides better short term kinematic and functional performance compared to those TKR's performed with ShapeMatch cutting guides modified to provide neutral overall limb alignment or with conventional instrumentation intended to achieve neutral overall limb alignment.
Time Frame: 6 months
Population: Early study termination resulted in limited availability of data for analysis to provide robust, meaningful results. Therefore the fluoroscopic data sets of the Neutral Overall Limb Alignment and Conventional Limb Alignment groups were combined and compared with the Kinematic Alignment group.
Measure: Mean (Standard Deviation); unit: Degrees
Arm/Group | Triathlon® CR/Kinematic Alignment | Triathlon® CR/Neutral Overall Limb Alignment | Triathlon® CR/Conventional Limb Alignment
Number analyzed (Participants) | 6 | 11 | 0
Degrees
  Contact Point Rotation (CPR) Stair Climbing | 7.3 (3.5) | 8.2 (3.2) |
  CPR Chair Rising | 12.6 (2.6) | 10.2 (3.7) |
  CPR Extension-Against-Gravity | 12.5 (4.2) | 8.8 (5.3) |

2. Secondary Outcome: Investigation of Clinical Performance and Patient Outcome With the Get-up and go Test
Description: Get-up-and-go test uses the time that a person takes to rise from a chair, walk three meters, turn around, walk back to the chair, and sit down.
  One source suggests that scores of ten seconds or less indicate normal mobility, 11 - 20 seconds are within normal limits for frail elderly and disabled patients, and greater than 20 seconds means the person needs assistance outside and indicates further examination and intervention. A score of 30 seconds or more suggests that the person may be prone to falls.
Time Frame: 1 year
Population: Due to early study termination, there was limited data available for analysis and therefore insufficient power to provide robust, meaningful results for our primary or secondary analysis.
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | Triathlon® CR/Kinematic Alignment | Triathlon® CR/Neutral Overall Limb Alignment | Triathlon® CR/Conventional Limb Alignment
Number analyzed (Participants) | 15 | 7 | 14
seconds | 5 (2.9) | 6 (2.8) | 7 (2.5)

3. Secondary Outcome: Investigation of Clinical Performance and Patient Outcome With the Knee Injury and Osteoarthritis Outcome Score (KOOS) Patient Questionnaire.
Description: KOOS consists of 5 subscales: Pain, other symptoms, function in daily living , function in sport and recreation and knee related quality of life (QOL). The previous week is the time period considered when answering the questions. Standardized answer options are given (5 Likert boxes) and each question is assigned a score from 0 to 4. A normalized score (100 indicating no symptoms and 0 indicating extreme symptoms).
Time Frame: 1 year follow-up
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Triathlon® CR/Neutral Overall Limb Alignment | Triathlon® CR/Kinematic Alignment | Triathlon® CR/Conventional Limb Alignment
Number analyzed (Participants) | 7 | 15 | 14
units on a scale
  Symptoms | 75 (20.0) | 84 (11.6) | 82 (11.7)
  Pain | 88 (13.7) | 91 (12.7) | 87 (15.2)
  Daily Living Activities | 89 (10.6) | 92 (8.9) | 86 (13.4)
  Sport/Recreation | 47 (25.1) | 58 (28.3) | 64 (27.3)
  Quality of Life | 89 (13.8) | 82 (19.9) | 76 (21.6)

4. Secondary Outcome: Investigation of Clinical Performance and Patient Outcome With the Forgotten Joint Score (FJS) Patient Questionnaire.
Description: The FJS consists of 12 questions and focuses on the patients' awareness of their joint replacement during a range of day to day and recreational activities. The score has a range of 0-100. High scores indicate good outcome, i.e., a high degree of being able to forget about the affected joint in daily life.
Time Frame: 1 year follow-up
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Triathlon® CR/Kinematic Alignment | Triathlon® CR/Neutral Overall Limb Alignment | Triathlon® CR/Conventional Limb Alignment
Number analyzed (Participants) | 15 | 7 | 14
units on a scale | 66 (32.1) | 82 (15.6) | 69 (27.7)

5. Secondary Outcome: Investigation of Clinical Performance and Patient Outcome With the EuroQuol-5 Dimension Health Questionnaire (EQ-5D).
Description: The EQ-5D index has an upper bound equal to 1 that indicates full health (indicated by "no problem" in all domains), whereas 0 represents death. Negative values are allowed, and the lower bound varies depending on country-specific value set used. UK time Trade Off (UKTTO) indicates the patient status compared to the normal state of the UK population.
Time Frame: 1 year follow-up
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Triathlon® CR/Kinematic Alignment | Triathlon® CR/Neutral Overall Limb Alignment | Triathlon® CR/Conventional Limb Alignment
Number analyzed (Participants) | 15 | 7 | 14
units on a scale | 0.9 (0.14) | 0.8 (0.12) | 0.9 (0.12)

6. Secondary Outcome: Investigation of Clinical Performance and Patient Outcome With the Short Form - 36 Health Survey (SF-36).
Description: The SF-36 Health Survey is a 36-item patient completed questionnaire to measure general health and well-being. It includes a physical and mental status component score; each ranging from 0-100. Low values represent a poor health state and high values represent a good health state.
Time Frame: 1 year follow-up
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Triathlon® CR/Kinematic Alignment | Triathlon® CR/Neutral Overall Limb Alignment | Triathlon® CR/Conventional Limb Alignment
Number analyzed (Participants) | 15 | 7 | 14
units on a scale
  Physikal Function | 51 (4.4) | 47 (6.3) | 48 (6.4)
  Role Physical | 50 (7.0) | 48 (11.3) | 48 (7.9)
  Bodily Pain | 54 (9.5) | 46 (11.5) | 49 (8.1)
  General Health | 51 (6.7) | 50 (6.1) | 54 (7.4)
  Vitality | 57 (9.3) | 54 (7.8) | 57 (9.1)
  Social Functioning | 50 (10.0) | 52 (7.9) | 53 (5.7)
  Role Emotional | 50 (6.5) | 45 (6.6) | 49 (10.2)
  Mental Health | 53 (7.0) | 50 (9.4) | 51 (11.5)

7. Secondary Outcome: Assessment of Better Performance of TKR Using a Kinematic Aligned ShapeMatch Cutting Guide by Functional Evaluation With Knee Society Score (KSS).
Description: The Knee Society Clinical Rating System is comprised of two distinct sub-scores: one for pain, Range of motion (ROM) and joint stability, and one for functional parameters. Sub-scores range from a potential minimum score of 0 to a maximum score of 100 points. Although the specific scores are not distinguished as "excellent," "good," "fair," or "poor," a higher value represents a better outcome.
Time Frame: 1 year follow-up
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Triathlon® CR/Kinematic Alignment | Triathlon® CR/Neutral Overall Limb Alignment | Triathlon® CR/Conventional Limb Alignment
Number analyzed (Participants) | 15 | 7 | 14
units on a scale
  Assessment Score | 87 (11.2) | 84 (16.1) | 82 (8.9)
  Function Score | 91 (17.7) | 89 (14.6) | 97 (4.7)

ADVERSE EVENTS:
Arm/Group | Triathlon® CR/Kinematic Alignment | Triathlon® CR/Neutral Overall Limb Alignment | Triathlon® CR/Conventional Limb Alignment
Serious Adverse Events (participants affected / at risk) | 1/15 | 4/11 | 2/18
Other Adverse Events (participants affected / at risk) | 0/15 | 0/11 | 0/18
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Triathlon® CR/Kinematic Alignment (N=15) | Triathlon® CR/Neutral Overall Limb Alignment (N=11) | Triathlon® CR/Conventional Limb Alignment (N=18)
Flexion deficit (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Instability (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Mammary Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Prostatic cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)

LIMITATIONS AND CAVEATS:
Due to early study termination, there was limited data available for analysis and therefore insufficient power to provide robust, meaningful results for our primary or secondary analysis.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less